CLINICAL TRIAL: NCT05545293
Title: Safety and Feasibility of Double-Stapling End-to-End Gastroduodenostomy Billroth-I Anastomosis in Laparoscopy-Assisted Surgery for Locally Advanced Distal Gastric Cancers: A Prospective Cohort Study
Brief Title: Prospective Study on Double-Stapling End-to-End Gastroduodenostomy Billroth-I Anastomosis in Laparoscopy-Assisted Surgery for Locally Advanced Distal Gastric Cancers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yong Zhou, Clinical Professor, West China Hospital
Other Study IDs: YZhou
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Advanced Gastric Carcinoma
Keywords: anastomotic leakage; laparoscopy-assisted surgery; double-stapling end-to-end gastroduodenostomy; Billroth-I anastomosis; anastomotic stenosis
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to explore the clinical application value of Double-Stapling End-to-End Gastroduodenostomy Billroth-I Anastomosis in Laparoscopy-Assisted Surgery for Locally Advanced Distal Gastric Cancers.

DETAILED DESCRIPTION:
As one of the core contents of gastric cancer surgery, the choice of digestive tract reconstruction method has always been the focus of clinical research in gastric cancer surgery. There are many alternative methods of digestive tract reconstruction at present, but there is no absolute superiority among various reconstruction methods. According to the individual characteristics of patients, the selection of appropriate digestive tract reconstruction methods should be an important direction in the future research field of digestive tract reconstruction.

There are many methods of digestive tract reconstruction in distal gastrectomy, including Billroth-I anastomosis, Billroth-II anastomosis and Roux-en-Y anastomosis. However, the standard method of reconstruction after distal subtotal gastrectomy does not reach a consensus. According to Korean Practice Guideline for Gastric Cancer 2018, gastroduodenostomy and gastrojejunal anastomosis are recommended after distal subtotal gastrectomy for middle-low gastric cancer, but the priority of different surgical procedures is not clarified. The conclusion is that there is no significant difference between the Billroth-I, Billroth-II and Roux-en-Y in postoperative quality of life, nutritional status and long-term prognosis of patients. Roux-en-Y anastomosis has a lower incidence of bile reflux, but a higher incidence of delayed gastric emptying compared with Billroth-I and Billroth-II. Similarly, the Japanese gastric cancer treatment guidelines in 2018 did not specify the priority of reconstruction methods after distal gastrectomy. In China, the 2022 CSCO guidelines for the diagnosis and treatment of gastric cancer also did not specify the priority of reconstruction methods, pointing out that alternative reconstruction methods include Billroth-I, Billroth-II combine with Braun anastomosis, Roux-en-Y anastomosis, and jejunal interposition. However, the number of alternative methods indicates that no ideal reconstruction method has absolute advantages. Therefore, in clinical practice, the specific choice of digestive tract reconstruction method often needs to be determined by considering many factors, including the location of the primary tumor, tumor stage, lymph node condition, anatomical variation and patient's economic situation, etc., which are important factors affecting the choice of digestive tract reconstruction method.

With the development of laparoscopic technique in recent years, totally laparoscopic digestive tract reconstruction has become a hot spot in the surgical treatment of gastric cancer. Laparoscopic digestive tract reconstruction has smaller incision and less trauma, which is a higher-level laparoscopic surgery pursued by surgeons. However, for patients undergoing radical gastrectomy for distal gastric cancer, totally laparoscopic distal gastroduodenal anastomosis is technically difficult. Delta anastomosis was proposed by Professor Kannaya in Japan in 2002. In this technique, the functional end to end anastomosis of the posterior wall of the remnant gastroduodenal was completed by using endoscopic linear staplers under totally laparoscopy, and the suture nails inside the anastomosis were triangular. It is a widely used functional end to end anastomosis of remnant gastroduodenum after distal gastrectomy under totally laparoscopic surgery. However, because of the operation in the duodenum and stomach from broken should meet the requirements of R0 resection of tumor, proper anastomotic tension, and blood supply of free longer duodenal stump, its restrictive factors, poor controllability, security is still not widely recognized, it can only be carried out in centers with rich experience in laparoscopic surgery, and it is more suitable for early cases of gastric Antrum.

In 2016, Professor Changming Huang found that modified Delta anastomosis is safe and feasible in early gastric cancer, but caution is still needed for locally advanced gastric cancer, its incidence of postoperative complications and anastomotic leakage was significantly higher than that of laparoscopic-assisted Billroth-I anastomosis.

In 1995, Oka et al. reported the use of circular stapler for functional end to end anastomosis of remnant gastroduodenum in open distal gastric cancer radical resection. In 2004, they reported the results of 221 cases, showing that this anastomosis was clinically safe and reliable. In 2007, Yang et al. in Korea confirmed that functional end to end anastomosis was safe and feasible in 933 cases of distal gastric cancer, with similar short-term outcomes compared with Billroth-II anastomosis. However, the clinical staging of gastric cancer patients in Japan and Korea is mainly early stage, but in China, the clinical staging of gastric cancer patients is mostly advanced stage.

In conclusion, traditional Billroth-I end-to-side anastomosis and Delta anastomosis require an additional residual gastric tissue of at least 3cm. In addition, the safe margin of the broken end of advanced gastric cancer requires a distance of at least 3-5 cm from the tumor, which often leads to higher anastomotic tension and significantly increases the risk of anastomotic leakage. Therefore, we propose a new technique for gastrointestinal reconstruction in laparoscopic distal radical gastrectomy in locally advanced gastric cancer: Double-Stapling End-to-End Gastroduodenostomy Billroth-I Anastomosis in Laparoscopy-Assisted Surgery. After previous practice, this anastomotic method can not only ensure a safe surgical margin, but also retain more residual stomach, so as to effectively solve the problem of anastomotic tension. It is a safe, simple, physiological and economic anastomotic method.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to years (including 18 and 85years old)
* Pathological diagnosis of primary focus is gastric adenocarcinoma made by endoscopic biopsy (papillary, tubular, mucinous, signet ring cell, poorly differentiated)
* cT1-4a, N+/-, M0 at preoperative evaluation
* No peritoneal metastasis or other distant metastases of gastric carcinoma (affirmed by laparoscopic surgery and related imaging examinations)
* Expected curative resection through laparoscopic distal gastrectomy with D2 lymphadenectomy (include multiple primary lower gastric adenocarcinoma)
* Performance status of 0 or 1 on Eastern Cooperative Oncology Group scale (ECOG)
* Preoperative American Society of Anesthesiology score (ASA) classⅠ, Ⅱ or Ⅲ
* Major organs are functioning normally:

blood routine test (No blood transfusions in the last 14 days): HB≥90g/L, ANC≥1.5×109/L, PLT≥80×109/L blood biochemical examination: BIL<1.5× upper limit of normal (ULN), ALT and AST<2.5×ULN, Crea≤1×ULN.

- The subject is willing to participate in this clinical trail

Exclusion Criteria:

* History of previous upper abdominal surgery (include ESD/EMR, except laparoscopic cholecystectomy)
* History of acute pancreatitis
* Regional fusion of enlarged lymph nodes by preoperative imaging (maximum diameter >3cm)
* History of other malignant disease within past five years
* History of unstable angina, myocardial infarction, cerebral infraction, or cerebral hemorrhage within past six months
* History of continuous systematic corticosteroids therapy within past one month
* Requirement of simultaneous surgery for other disease
* Emergency surgery due to complication (bleeding, or perforation) caused by gastric cancer
* FEV1<50% of predicted values by pulmonary function test
* Women during pregnancy or breast-feeding
* Severe mental disorder
* Participating in other clinical studies simultaneously
* Refusing to sign the informed consent for the study
* Peritoneal implant or other distant metastases by intraoperative exploration
* Unresectable due to tumor reasons by intraoperative exploration
* Distal gastric cancer surgery cannot be performed after intraoperative exploration
* Duodenal bulb has been invaded by tumor or gastroduodenostomy cannot be performed due to additional surgical resection cause by positive intraoperative frozen margin

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients enrolled in this study would undergo double-stapling end-to-end gastroduodenostomy Billroth-I anastomosis in laparoscopy-assisted surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-14 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Anastomotic complications | up to 1-30 Days after surgery
  The anastomotic complications are defined as the event observed within 30 days after surgery, including anastomotic stenosis, anastomotic bleeding, and anastomotic leakage.
Intraoperative situation | on the day of surgery
  Operation time, anastomotic reconstruction time, operative blood loss, completed proportion of laparoscopic surgery, positive rate of Intraoperative frozen margin pathology, anastomotic tension, the distance between proximal and distal of resection margin, the incidence of complication in surgery are used to access the intraoperative situation.
Postoperative nutritional status and quality of life | up to 1-30 Days after surgery
  The variation of weight, cholesterol and albumin on postoperative 30 days are used to access the postoperative nutritional status and quality of life.

SECONDARY OUTCOMES:
Length of hospital stay | up to 1-30 Days after surgery
  The time between end of surgery and written discharge ticket
Cost of hospitalization | up to 1-30 Days after hospital admission
  The fees paid during the course of this hospitalization
Other postoperative complications | up to 1-30 Days after surgery
  Other postoperative complications are defined as events other than anastomotic complications occurring within 30 days after surgery.
Postoperative intestinal function recovery time | up to 1-6 Days after surgery
  The time between end of surgery and first bowel movement

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nishizaki D, Ganeko R, Hoshino N, Hida K, Obama K, Furukawa TA, Sakai Y, Watanabe N. Roux-en-Y versus Billroth-I reconstruction after distal gastrectomy for gastric cancer. Cochrane Database Syst Rev. 2021 Sep 15;9(9):CD012998. doi: 10.1002/14651858.CD012998.pub2. PMID 34523717
- [Result] Japanese Gastric Cancer Association. Japanese gastric cancer treatment guidelines 2018 (5th edition). Gastric Cancer. 2021 Jan;24(1):1-21. doi: 10.1007/s10120-020-01042-y. Epub 2020 Feb 14. No abstract available. PMID 32060757
- [Result] Cai Z, Zhou Y, Wang C, Yin Y, Yin Y, Shen C, Yin X, Chen Z, Zhang B. Optimal reconstruction methods after distal gastrectomy for gastric cancer: A systematic review and network meta-analysis. Medicine (Baltimore). 2018 May;97(20):e10823. doi: 10.1097/MD.0000000000010823. PMID 29768387
- [Result] Jin HE, Kim MS, Lee CM, Park JH, Choi CI, Lee HH, Min JS, Jee YS, Oh J, Chae H, Choi SI, Lee YT, Kim JH, Huang H, Park S. Meta-analysis and systematic review on laparoscopic-assisted distal gastrectomy (LADG) and totally laparoscopic distal gastrectomy (TLDG) for gastric cancer: Preliminary study for a multicenter prospective KLASS07 trial. Eur J Surg Oncol. 2019 Dec;45(12):2231-2240. doi: 10.1016/j.ejso.2019.06.030. Epub 2019 Jun 22. PMID 31262598
- [Result] Kanaya S, Gomi T, Momoi H, Tamaki N, Isobe H, Katayama T, Wada Y, Ohtoshi M. Delta-shaped anastomosis in totally laparoscopic Billroth I gastrectomy: new technique of intraabdominal gastroduodenostomy. J Am Coll Surg. 2002 Aug;195(2):284-7. doi: 10.1016/s1072-7515(02)01239-5. No abstract available. PMID 12168979
- [Result] Lin M, Zheng CH, Huang CM, Li P, Xie JW, Wang JB, Lin JX, Lu J, Chen QY, Cao LL, Tu RH. Totally laparoscopic versus laparoscopy-assisted Billroth-I anastomosis for gastric cancer: a case-control and case-matched study. Surg Endosc. 2016 Dec;30(12):5245-5254. doi: 10.1007/s00464-016-4872-3. Epub 2016 Mar 23. PMID 27008576
- [Result] Oka M, Maeda Y, Ueno T, Iizuka N, Abe T, Yamamoto K, Ogura Y, Masaki Y, Suzuki T. A hemi-double stapling method to create the Billroth-I anastomosis using a detachable device. J Am Coll Surg. 1995 Oct;181(4):366-8. No abstract available. PMID 7551332
- [Result] Kuwabara Y, Shinoda N, Sato A, Kimura M, Ishiguro H, Sugiura H, Tanaka T, Ando T, Fujii Y, Fujii Y. Billroth I gastroduodenostomy using a hemi-double stapling technique. J Am Coll Surg. 2004 Apr;198(4):670-2. doi: 10.1016/j.jamcollsurg.2003.11.016. No abstract available. PMID 15051021
- [Result] Park SH, Kang MJ, Yun EH, Jung KW. Epidemiology of Gastric Cancer in Korea: Trends in Incidence and Survival Based on Korea Central Cancer Registry Data (1999-2019). J Gastric Cancer. 2022 Jul;22(3):160-168. doi: 10.5230/jgc.2022.22.e21. PMID 35938363
- [Result] Yang HK, Lee HJ, Ahn HS, Yoo MW, Lee IK, Lee KU. Safety of modified double-stapling end-to-end gastroduodenostomy in distal subtotal gastrectomy. J Surg Oncol. 2007 Dec 1;96(7):624-9. doi: 10.1002/jso.20883. PMID 17708549